CLINICAL TRIAL: NCT04835571
Title: CARotid Mri of Atherosclerosis
Acronym: CARMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other); Region Jönköping County (Other Government); FORSS, Forskningsrådet i Sydöstra Sverige (Unknown)
Responsible Party: Principal Investigator, Ebo De Muinck, Professor Ebo de Muinck, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 756191
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Carotid Stenosis; Carotid Artery Plaque; Carotid Atherosclerosis
Keywords: Carotid stenosis; Cardiovascular MRI; Atherosclerotic plaque
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases; Plaque, Atherosclerotic

STUDY DESIGN:
Intervention Model Description: Single group, repeated measures design. The treatment is
Oversight: Data Monitoring Committee: No

ARMS (1):
- CARMA study participants (Experimental): All patients in the study are in the same treatment arm: all were treated for 12 months according to routine care and international guidelines for cardiovascular disease prevention in patients with very high cardiovascular risk. Through study physicians patients received an individual assessment and optimized cardiovascular risk management, including life style advice and adjustments in their medical preventive treatment, based on drugs used in standard care (eg. lipid lowering medication, anti-hypertensive-treatment, anti-thrombotic treatment). All treatment goals were set in accordance with current guidelines at the time for study participation.
  Interventions: Other: Optimization of cardiovascular risk management

INTERVENTIONS:
Other: Optimization of cardiovascular risk management — Treatment goals were set according to current guidelines (Perk et al. Eur Guidelines on CVD prevention in clinical practice (2012). Eur heart J. 2012;33(13):1635-701):
  * blood pressure <140/90 mmHg
  * Tot cholesterol <5 mmol/l
  * LDL <1,8 mmol/l
  * Waist circumference: men <94 cm, women <80 cm
  * BMI <25 kg/m2
  * HbA1c without diabetes mellitus <42 mmol/mol, HbA1c with diabetes mellitus <52 mmol/mol
  * Antithrombotic treatment (or anticoagulants, if indicated)
  * Physical activity 30 min/day, 5 days/week, alternatively high-intensity training at least15 min/day, 5 days/week or a combination of the two.
  * Healthy diet, including low levels of saturated fats, high intake of vegetables, fruits, whole-grain and fish
  * Smoking cessation
  * Low alcohol consumption
  Patients were encouraged to follow the above recommendations through support of the study physicians, who made individual assessments of all patients and adjusted ongoing medical treatment to reach treatment targets.

SUMMARY:
In the entire world most people die from cardiovascular disease. Death is primarily from myocardial infarction (MI) and stroke which are most often caused by rupture of atherosclerotic plaques. Patients with high-grade, i.e. ≥ 70% carotid artery stenosis are at especially high risk. Magnetic Resonance Imaging (MRI) studies show that two features inside plaques that are associated with the risk of plaque rupture and subsequent cardiovascular events are: lipid rich necrotic core (LRNC) and intraplaque hemorrhage (IPH).

MRI studies on carotid artery plaques typically relies on proton-density-weighted fast-spin echo, blood-suppressed T1- and T2-weighted gradient-echo sequences. The end-result is nonquantitative measures, where plaque features are identified due to their relative signal intensity. To address these problems of non-specificity, we developed a quantitative MRI (qMRI) technique based on Dixon sequences.

The study intention is to enable in-depth analysis of plaque features and their relation to clinical data. For example there is an insufficient understanding of associations between lipid biomarkers and plaque contents. Our hypothesis is that we can identify quantitative changes in both plaque and lipid biomarkers after one year of optimized cardiovascular risk management (including treatment with lipid lowering drugs), and establish if there is any associations between these features. Because there is a well-established link between systemic inflammation and the presence of atherosclerotic plaques we will also study the relationship between LRNC and IPH as measured by qMRI versus circulating markers of inflammation.

Method: Patients with known carotid stenosis are invited for a baseline visit and a 1-year follow up visit. The study visits include clinical assessment, blood tests, patient interview and magnetic resonance imaging of the carotid arteries. All participants are offered optimized cardiovascular risk management through the individual assessment by the study physicians.

DETAILED DESCRIPTION:
Regarding quality assurance plans that address data validation and registry procedures, the current study is a single centre investigator-initiated study and therefore there are no plans for site monitoring and auditing. The reliability and validity of the MRI data has been previously confirmed with comparison to 3D histology data (Koppal et al. Quantitative fat and R2* mapping in vivo to measure lipid-rich necrotic core and intraplaque hemorrhage in carotid atherosclerosis. Magn Reson Med. 2017;78(1):285-96.).

Concerning data checks, intraobserver reliability regarding baseline and follow-up measurements will be ascertained (Intraclass Correlation Coefficients (ICC), Bland Altman).

Data is collected from patient medical records (electronic), dedicated study record forms (paper) and clinical assessments, resulting in quantitative measures. These external data sources are transferred into a study database.

The current study is a clinical study, using only clinically validated laboratory parameters. The source of the lab values and their normal ranges is the electronic patient record. The normal ranges have been established by the clinical chemistry and haematology laboratories at Linköping University Hospital. Clinical diagnosis and procedures are recorded using the International Classification of Diseases (ICD) classification.

The study was approved by the Swedish Ethical Review Authority (approval nr: 2016-441-31) and performed in accordance with the Declaration of Helsinki. Written informed consent has been obtained from all study participants.

Patients are selected based on duplex ultrasound criteria established for the European Carotid Surgery Trial. A cut-off at doppler flow velocity has been used to identify eligible patients and after considering inclusion and exclusion criteria patients have been contacted by the study clinicians dr Elin Good or dr Ebo de Muinck for recruitment. Any registration for adverse events follows the same procedures as in routine care.

Sample size assessment was based on results from previous studies in relation to our primary outcome variables. For example, one study with 24 patients and a follow-up time of three months experienced a significant reduction of lipid rich necrotic core, using magnetic resonance imaging (Alkhalil et al. T2 mapping MRI technique quantifies carotid plaque lipid, and its depletion after statin initiation, following acute myocardial infarction. Atherosclerosis. 2018;279:100-6.). Therefore, we aimed to include 50 patients who have completed both baseline and follow-up, and the follow-up time was set to 12 months.

Our plan for missing data in situations where variables are missing, unavailable, non-reported, uninterpretable etc is to not exclude the study participant, in order to avoid bias. For example, in cases where the imaging data from one patient is lost, we will still use the remaining clinical data from that patient if the patient has been included in the study.

Regarding Statistical analysis, SPSS Statistics 26 (International Business Machines Corporation, New York, NY, USA) is used for statistical analysis. Continuous variables are summarized as mean ± standard deviation (SD). To address the primary objectives (the strength of the association between fat fraction (FF) and R2*) Pearson correlation coefficient is used, and Paired-samples T test is used for analysing changes in quantitative values between baseline and follow-up.

Intra-observer repeatability measurements were calculated using ICC. For ICC evaluation we used two-way random effect models, checking for absolute agreement, average measures presented.

ELIGIBILITY:
Inclusion Criteria:

- Carotid plaques with a cut-off at doppler flow velocity ≥ 1.3 m/sec at a Doppler angle of 50-60°, which corresponds to a ≥ 50% stenosis according to these criteria.

Exclusion Criteria:

* Performed or planned carotid surgery
* Carotid occlusion
* Renal failure (GFR <45 ml/h)
* Inflammatory diseases, anti-inflammatory treatment or malignancies
* Stroke <30 days before admission
* Co-morbidities that disable informed consent or participation in the study investigations (e.g. contraindications for MRI)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in fat fraction (FF) and R2* in relation to changes in plasma lipoproteins. | Baseline - 1-year follow up
  FF, Fat Fraction. Measured by Dixon MRI sequences, quantitatively corresponding to lipid rich necrotic core. R2* (= 1/T2*) is the rate of signal loss, it can be viewed as a measure for the presence of (heme) iron. As we have shown in a previous study, it correlates to the extent of intraplaque hemorrhage.

SECONDARY OUTCOMES:
Changes in fat fraction (FF) and R2* in relation to changes in inflammatory lymphocyte subtypes | Baseline - 1-year follow up
  For FF and R2*, see above. Inflammatory lymphocytes subtypes are measured using flow cytometry, with focus on lymphocyte T cell subtypes and Natural Killer cells.

CONTACTS AND LOCATIONS:
Overall Officials: Ebo de Muinck, Professor, Principal Investigator — Linkoeping University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koppal S, Warntjes M, Swann J, Dyverfeldt P, Kihlberg J, Moreno R, Magee D, Roberts N, Zachrisson H, Forssell C, Lanne T, Treanor D, de Muinck ED. Quantitative fat and R2* mapping in vivo to measure lipid-rich necrotic core and intraplaque hemorrhage in carotid atherosclerosis. Magn Reson Med. 2017 Jul;78(1):285-296. doi: 10.1002/mrm.26359. Epub 2016 Aug 11. PMID 27510300
- [Background] Good E, Lanne T, Wilhelm E, Perk J, Jaarsma T, de Muinck E. High-grade carotid artery stenosis: A forgotten area in cardiovascular risk management. Eur J Prev Cardiol. 2016 Sep;23(13):1453-60. doi: 10.1177/2047487316632629. Epub 2016 Feb 15. PMID 26879568
- [Derived] Good E, Akerman L, Nystrom S, Jonasson L, Ernerudh J, de Muinck E. Changes in natural killer and T lymphocyte phenotypes in response to cardiovascular risk management. Sci Rep. 2023 Nov 27;13(1):20810. doi: 10.1038/s41598-023-48111-7. PMID 38012327